CLINICAL TRIAL: NCT07370454
Title: Clinical Evaluation of the Xpert Hemorrhagic Fever Test Using Clinical Specimens and Contrived Samples on the GeneXpert Edge X System
Brief Title: Xpert® Hemorrhagic Fever on the GeneXpert® Edge X System
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Responsible Party: Sponsor
Other Study IDs: P259C
Record Dates: First submitted 2025-10-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fevers, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Capillary and venous whole blood specimens: whole blood specimens from individuals asymptomatic or symptomatic of fever
  Interventions: Diagnostic Test: Xpert Hemorrhagic Fever test

INTERVENTIONS:
Diagnostic Test: Xpert Hemorrhagic Fever test — Detection and identification of RNA from multiple viruses from whole blood specimens

SUMMARY:
A multi-site observation study that was conducted a geographically diverse sites across the United States

DETAILED DESCRIPTION:
Capillary and venous whole blood specimens were prospectively collected from consented individuals symptomatic or asymptomatic of fever

ELIGIBILITY:
Inclusion Criteria:

* Capillary and venous whole blood specimens from blood donors who symptomatic for fever lasting ≤ 10 days OR asymptomatic for fever
* Whole blood specimens collected in EDTA specimens collection devices only

Exclusion Criteria:

* Any whole blood specimens from blood donors vaccinated with a Hemorrhagic Fever live virus vaccine within the past 28 days
* Any whole blood specimen that were previously enrolled
* Any whole blood specimens not collected according to the manufacturer's instructions

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Whole blood specimens collected from blood donors symptomatic or asymptomatic of fever
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Clinical performance comparing Xpert Hemorrhagic Fever to known status of specimens | Clinical Performance assessed in specimens collected at Baseline
  Xpert test compared to expected status

CONTACTS AND LOCATIONS:
Locations (1):
- USAMRIID, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No